CLINICAL TRIAL: NCT04817176
Title: Pilot Trial of an Motivational Interviewing-Cognitive Behavioral Therapy Ketogenic Nutrition Adherence Program for Older Adults
Brief Title: MI-CBT Adherence Program for Lifestyle Interventions in Older Adults
Acronym: MI-CBT KNAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Julia Sheffler, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1KL2TROO1429; 1KL2TROO1429 (Other Grant/Funding Number: NIH NCATS); P30AG059297 (NIH)
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Mild Cognitive Impairment; Adherence, Patient; Ketosis
MeSH Terms: conditions — Cognitive Dysfunction; Patient Compliance; Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI-CBT KNA Program (Experimental): The program is a 6-week group, telehealth intervention for older adults with possible MCI. The intervention uses Motivational interviewing and cognitive behavioral therapy strategies to enhance motivation and help participants overcome personal obstacles to following health-behavior recommendations. Specifically, the program examines the use of a Mediterranean ketogenic type of nutrition to target mild cognitive impairment. The intervention is designed to disseminate practical information to help older adults learn how to incorporate healthy Mediterranean ketogenic nutrition into their lifestyle.
  Interventions: Behavioral: Motivational Interviewing-Cognitive Behavioral Therapy Ketogenic Nutrition Adherence Program
- KN Information-Only Program (Active Comparator): 6-week group, telehealth intervention for older adults. The intervention is designed to disseminate practical information to help older adults learn how to incorporate healthy Mediterranean ketogenic nutrition into their lifestyle.
  Interventions: Other: Ketogenic Nutrition Program

INTERVENTIONS:
Behavioral: Motivational Interviewing-Cognitive Behavioral Therapy Ketogenic Nutrition Adherence Program — Experimental Arm: The program is a 6-week group, telehealth intervention for older adults with possible MCI. The intervention uses Motivational interviewing and cognitive behavioral therapy strategies to enhance motivation and help participants overcome personal obstacles to following health-behavior recommendations. Specifically, the program examines the use of a Mediterranean ketogenic type of nutrition to target mild cognitive impairment. The intervention is designed to disseminate practical information to help older adults learn how to incorporate healthy Mediterranean ketogenic nutrition into their lifestyle.
  Arms: MI-CBT KNA Program
Other: Ketogenic Nutrition Program — Active Comparator Arm: 6-week group, telehealth intervention for older adults. The intervention is designed to disseminate practical information to help older adults learn how to incorporate healthy Mediterranean ketogenic nutrition into their lifestyle.
  Other Names: KN Information-Only
  Arms: KN Information-Only Program

SUMMARY:
Objective 1:

Assess feasibility and acceptability of all protocol components of a pilot trial testing a 6-week telehealth Mediterranean ketogenic nutrition adherence (KNA) program using motivational interviewing and cognitive behavioral strategies (MI-CBT) compared to a KN information only group for older adults with mild cognitive impairment (MCI) to prepare for a full-scale trial.

Specifically, the investigators will examine the feasibility of the recruitment, retention, assessment, and intervention delivery methods.

The investigators hypothesize that:

1. The study protocol will result in high patient retention (90%) and patient attendance of intervention sessions (80%), and
2. A centralized MI-CBT telehealth delivery approach will be associated with high intervention acceptability ratings from patients.

Objective 2:

Assess signal of initial effect of the KNA program on important clinical outcomes and adherence relative to a KN information-only condition.

The investigators hypothesize that patients in the KNA condition, relative to the KN-only condition, will show:

1. higher rates of clinically significant improvements on the RBANS total scale scores, improvements in daily functioning (FSQ), and decreases in patient CAIDE risk score( (Cardiovascular Risk Factors, Aging, and Incidence of Dementia), and
2. improved adherence to KN, as evidenced by higher levels of measurable urine ketones in the KNA condition compared to the KN-only condition.

DETAILED DESCRIPTION:
Preparation. During the first 6 months of the study, the investigators will work closely with key stakeholders (i.e., clinic director, practice manager, and nurse practitioner) in the Florida State University (FSU) SeniorHealth clinic to coordinate initial contact with patients about the study. Initial contact will include posting flyers in the SeniorHealth clinic, handing out flyers during appointments, and emailing flyers or calling patients who have consented to be contacted about FSU research studies (a consent process, which is completed as part of the normal SeniorHealth intake packet), posting flyers in the Westminster Oaks monthly newsletter, and patients will be able to fill out a contact card with their name, phone number, and email that will be placed in a locked "drop box" in the SeniorHealth clinic. A study team member will collect these cards weekly to enter into a secure screening waitlist. Patients may also discuss interest with their provider or contact the study team directly using the information on the study flyer, potential participants will be added to a secure screening waitlist, which will include only their name and phone number. This screening waitlist potential participant contact information will be stored in a password protected document. Contact information for potential participants will be destroyed for any participant who does not qualify and consent to remain in the study.

Screening phone call. After confirming interest in being contacted about the study, participants will be contacted by a member of the research team and screened for eligibility. This screening will include a telephone Montreal cognitive assessment (MoCA), sections 1 and 4 from the Functional Status Questionnaire (FSQ), a brief memory complaint scale, and self-reported height, weight, and age. Participants will also be asked to report any restrictive dietary or medical conditions that may make them unable to change their nutrition. This contact information will not be retained for future research purposes. All screened participants will be provided with a handout on healthy living designed in collaboration with the SeniorHealth physicians. If participants are eligible, then they will be sent an online consent form, which they will read and review telephonically with a member of the research team before signing. The study team will then complete a final eligibility check of the patient's EHR and review with the physician to confirm eligibility and ensure participant safety. Participants who are eligible and consent to participate will have screening data linked with other study data, in order to reduce redundancy in assessment measures.

Pre-intervention EHR data download (Time 0). The research team will extract and clean relevant EHR data on participants who consent to participate in the study. Data from EHR will be used to conduct a secondary eligibility screening to determine if there are any other major health conditions that will exclude participants from the study. Data will only include the minimum protected health information (PHI) necessary to complete the proposed study. Data from the EHR will include the following information only from appointments pertinent to the study: patients' problem/diagnostic list, medication list, patient vitals, metabolic panels, HbA1C, scores on recent cognitive and psychological assessments (i.e., MoCA, depression inventories), and relevant provider notes about a patient's cognitive functioning. Participants that are seen by FSU clinicians will be considered for the study and contacted by our team. Their EHR is maintained on Athena and thus all the information will be accessed from Athena. Clinic staff working for FSU will be responsible for screening their EHR and determining their eligibility for the study. These data will include the participants MoCA scores, the geriatric depression inventory (GDS), and FSQ scores or relevant qualitative data about their activities of daily living, and demographic characteristics. The study team will also include laboratory results that may be relevant to cognitive outcomes for secondary data analyses, including: HbA1c, glucose, potassium, blood pressure, and cholesterol. All laboratory data will be pulled from the EHR, and will not require additional bloodwork or labs to be completed by patient participants.

Baseline Assessment (Time 1). In addition to embedded EHR data, we are collecting additional data to evaluate the personal impacts of the intervention. This assessment will include: the Repeatable Battery of Neuropsychological Status (RBANS update - form A), the GDS, FSQ, and CAIDE risk score. This assessment will be completed using HIPAA Compliant Zoom.

Post-intervention Assessment (Time 2). Participants will complete this assessment in the final weeks of the program, in order to assess participants when they are in ketosis. Participants will be asked to return their ketone logs either electronically, reported over the phone, or via mail to the study PI. The research team will complete qualitative interviews with participants to collect information about barriers and facilitators to completing the program and adhering to KN. Participants will complete the RBANS update - Form B, the GDS, and FSQ, and the client satisfaction questionnaire . This assessment will be completed using HIPAA Compliant Zoom.

Post-intervention EHR data download and Provider Assessment (Time 3). Approximately six months post-intervention, we will complete a final data extraction from the EHR, which will include the same data as Time 0. Additionally, we will complete semi-structured interviews with the clinic providers to assess implementation barriers and facilitators. Providers will also complete quantitative measures on implementation acceptability (i.e., Modified version of the Assessment of Fit Scale for outpatient clinics).

Post-intervention Assessment (Time 4). Patient participants will complete this assessment approximately 3 months after completing the intervention program, in order to assess long-term maintenance. The research team will complete qualitative interviews with participants to collect information about barriers and facilitators to adhering to KN long-term. Participants will complete the RBANS Update - form C, the GDS, and FSQ. This assessment will be completed using HIPAA Compliant Zoom.

Intervention Description:

Using a centralized telehealth approach, the KNA program will consist of 6 weekly group meetings, which will take place via HIPAA-compliant Zoom. The group will be co-led by a clinical psychologist and a licensed nutritionist. Approximately half of each session will be devoted to providing nutrition information and half devoted to psychoeducation, MI activities, and CBT skills. Each group session will be recorded and rated by a trained clinician using a modified MI Coach Rating Scale to measure fidelity to MI-CBT strategies and reviewed with a recognized expert on MI and CBT. These recordings will be stored on a secure College of Medicine network drive and will only be used for the duration of the project and reviewed by the study team for quality control and intervention consistency. Any information from these recordings used for research purposes will be fully de-identified, with qualitative information transcribed and coded by the research team.

MI-CBT KNA Week 1:

The first group meeting will consist of a 1.5 hour informational and psychoeducational session to introduce participants to the purpose of the group, the ketogenic nutrition goals, and to the MI-CBT model of behavior change in relation to nutrition. Participants will be mailed a workbook that includes weekly goals, handouts on how to maintain KN, including daily recipes and food lists, as well as MI-CBT handouts and worksheets. Participants will be asked to slowly begin reducing daily net carbohydrate intake to 125g over the first week.

The study team will provide individualized recommendations for macronutrient intake based on the net carbohydrate weekly goal and participant health information (e.g., sex, weight, height, activity level). Participants will log macronutrient intake in their food logs in order to ensure that approximately 60% of their diet involves healthy fats (e.g., fish, avocado, olive oils), and to begin learning the general macronutrient content of foods they consume. Participants will have the option of completing these food longs online or using paper copies at home. The focus of these first meetings will be on nutritional education and helping participants identify relevant values, goals, and reasons for committing to make healthy changes.

MI-CBT KNA Weeks 2-4:

In 1-hour weekly meetings, participants will learn about the CBT model and relevant skills, with assigned homework. Based on feedback from the feasibility trial, the program will emphasize cognitive restructuring and problem-solving as primary skills, while handouts on additional techniques (e.g., distress tolerance, behavioral activation, mindfulness) will be provided as optional.

These skills will help participants identify health goals, manage triggers for unhealthy eating behaviors, and overcome external obstacles to healthy eating. MI will be employed throughout these sessions, through worksheets as well as reflective listening, summarizing, affirming, and open-ended questions from the group leaders. Participants will be instructed to gradually reduce their net carbohydrate intake across the first 3 weeks of the program in a step-wise fashion (i.e., 125g in week 1, 75g in week 2, 50g or less in week 3) in order to reduce possible adverse responses to the diet (e.g., GI distress, fatigue). Healthy fat intake is a core component of this program, and participants will be provided with ample instruction on ways to increase healthy fat intake while maintaining a healthy balance of macronutrients (e.g., 60% fat, 30% protein, 10% carbohydrates).

MI-CBT KNA Weeks 5-6:

In the final two sessions, the focus will shift to emphasize CBT skills practice, maintenance of goals, sustainment of progress, and social support. Participants will make maintenance plans, learn to manage slips, and continue practicing cognitive restructuring skills. The recommended net carbohydrate intake will be reduced to 20g or less these weeks, depending on individual ketone level and macronutrients.

KN-Only (Condition 2):

Participants assigned to the KN-only group will attend a 1.5-hour informational session as a group, which will provide comprehensive information about how to adhere to KN and how to track macronutrients, food intake, and ketone levels. Participants will be provided with the same participant workbook as the MI-CBT KNA group with informational handouts and KN recipes, but without the MI-CBT handouts. Participants will be asked to track food intake and daily ketone levels, and will be provided with the option of attending a weekly Zoom meeting where they may ask questions about KN and receive additional nutrition information as needed. These optional meetings will be offered for 6 weeks. The structure of this control condition will allow us to examine of the benefits that an MI-CBT group approach provides for increasing adherence to KN and retention in a KN program, compared to KN education only.

MODIFICATION: EHR data collection and recruitment through the Senior Health clinic were determined to not be feasible based on the available patient data. The protocol was updated prior to the intervention to include collection of health and biomarker data during in-person assessments in place of EHR data collection. Recruitment was extended to all eligible community and independent living older adults and was not restricted to patients at the senior health clinic.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-85 years
* Meets criteria for possible mild cognitive impairment
* Telephone MoCA Score of greater than 12
* Reports interest in participating in the described nutrition intervention
* English speaking
* Has internet access with video conferencing capability and access to a computer, iPad, or other tablet.

Exclusion Criteria:

* Major, unstable health or psychiatric conditions, including: Type 1 diabetes, major neurocognitive disorders, schizophrenia, bipolar I disorder, or active psychosis
* Under-weight based on BMI
* Prescribed medications that may interact with ability to adhere to KN, including: insulin, monoamine oxidase inhibitors (MAOIs), or immunosuppressants
* Deemed unable to provide consent based on telephone cognitive screener with a licensed psychologist.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia L Sheffler, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sheffler JL, Kiosses DN, He Z, Arjmandi BH, Akhavan NS, Klejc K, Naar S. Improving Adherence to a Mediterranean Ketogenic Nutrition Program for High-Risk Older Adults: A Pilot Randomized Trial. Nutrients. 2023 May 16;15(10):2329. doi: 10.3390/nu15102329. PMID 37242211
- [Derived] Klejc K, Cruz-Almeida Y, Sheffler JL. Addressing Pain Using a Mediterranean Ketogenic Nutrition Program in Older Adults with Mild Cognitive Impairment. J Pain Res. 2024 May 23;17:1867-1880. doi: 10.2147/JPR.S451236. eCollection 2024. PMID 38803693

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MI-CBT KNA Program | KN Information-Only Program
Started | 29 | 29
Completed | 26 | 24
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MI-CBT KNA Program | KN Information-Only Program | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.59 (6) | 73.24 (6.77) | 72.91 (6.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 25 | 21 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Retention in the clinical intervention as assessed by percent of attendance at the intervention groups
Time Frame: 6-weeks
Measure: Number; unit: percentage of participants
Arm/Group | MI-CBT KNA Program | KN Information-Only Program
Number analyzed (Participants) | 29 | 29
percentage of participants | 90.6 | 76.6

2. Primary Outcome: Acceptability
Description: Acceptability will be assessed using the Client Satisfaction Questionnaire - 8, item 1, rated 1 (poor) - 4 (excellent) (How would you rate the quality of service you received?).
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale (1-4)
Arm/Group | MI-CBT KNA Program | KN Information-Only Program
Number analyzed (Participants) | 26 | 24
units on a scale (1-4) | 3.65 (0.57) | 3.6 (0.50)

3. Primary Outcome: Ketosis (Adherence)
Description: Participants will show measurable levels of ketones using at-home urinalysis test strips by week 5 of the intervention, as evidenced by greater than trace amounts of ketones on the urine test strips (i.e., >5mg/dl).
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: 6-week average urine ketone levels mg/dl
Arm/Group | MI-CBT KNA Program | KN Information-Only Program
Number analyzed (Participants) | 25 | 24
6-week average urine ketone levels mg/dl | 17.32 (14.41) | 10.54 (0.089)

4. Other Pre Specified Outcome: Brief Pain Inventory, Pain Intensity Scale
Description: Pain intensity was measured using 4 items in the BPI with possible responses ranging from "0=No Pain" to "10=Pain as Bad as You Can Imagine." Items included pain experienced "at its worst in the last 24 hours" and "pain on average" which were used to measure the magnitude of pain experienced by participants. Pain intensity was calculated as the mean of the 4 items in the BPI with total scores ranging from 0-10 and higher scores indicating worse pain intensity. Changes in pain intensity was calculated by subtracting the baseline total pain intensity score from the 6-week pain intensity score, with a higher negative value indicating greater improvement in pain intensity over time
Time Frame: 6 weeks
Population: participants must report pain at screening to be included in analyses
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- MKNA: Full ICAN adherence program
- MKNE: Educational comparator group
Arm/Group | MKNA | MKNE
Number analyzed (Participants) | 9 | 11
score on a scale | -0.111 (1.4) | -0.159 (1.2)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | MI-CBT KNA Program | KN Information-Only Program
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT04817176/Prot_000.pdf